CLINICAL TRIAL: NCT05406726
Title: Mechanisms of Palmitoylethanolamide (PEA) to Alter Pain Sensitivity in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jennifer Klinedinst, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HP-00101407
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — palmidrol; maltodextrin

STUDY DESIGN:
Intervention Model Description: This is a crossover clinical trial where 10 participants will receive palmitoylethanolamide (PEA) dietary supplement for 6 weeks and 10 participants will receive placebo for six weeks. Then the following six weeks they will reverse.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will occur as to the order of receiving either PEA or placebo for the first six weeks, then the reverse for the following six weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- palmitoylethanolamide (PEA) (Experimental): Palmitoylethanolamide (PEA) is a lipid based endocannabinoid dietary supplement currently marketed.
  Interventions: Dietary Supplement: palmitoylethanolamide
- Placebo (Placebo Comparator): A similar size and shaped capsule containing maltodextrin will be used as a placebo comparator.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: palmitoylethanolamide — palmitoylethanolamide is an lipid based endocannabinoid naturally made by the body and is present in several common foods such as eggs
  Other Names: PEA
  Arms: palmitoylethanolamide (PEA)
Dietary Supplement: Placebo — a capsule filled only with maltodextrin will be used as a placebo
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
The purposes of this 1-year proof of feasibility and acceptability pilot study are twofold. First to determine if participants with knee osteoarthritis (KOA) will comply with taking palmitoylethanolamide (PEA) dietary supplement for 6 weeks and adhere to taking it as directed. Second is to gain preliminary data to elucidate mechanisms (protein signatures, inflammatory markers and neurobiological signaling pathways) by which PEA, a lipid-based endocannabinoid, works to alter pain sensitivity in adults with KOA. In the simplest terms possible, we need to provide evidence that PEA changes the protein signature in order to provide evidence to establish mechanism.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) affects nearly 30% of adults aged 60 years or older and causes significant pain and disability.1 Neurophysiological testing (quantitative sensory testing (QST)) demonstrates that KOA pain has both peripheral and central mechanisms, which vary by individual.2 Adults with central KOA pain tend to be resistant to traditional pain treatment and have substantial pain even after knee replacement surgery.3 There is a growing body of evidence to support the scientific premise that endocannabinoids and related molecules, in particular PEA, can improve KOA pain through anti-inflammatory and analgesic pathways.4,5 PEA has little or no known side effects and is safe for human consumption.6 However, there is little known regarding the specific mechanisms by which PEA works to relieve KOA pain or for whom it might work best. We will begin to address this mechanistic question in this pilot study, which will provide data regarding therapeutic strategies within the endocannabinoid system to reduce KOA pain. The National Academies of Science, Engineering and Medicine report on the Health Effects of Cannabis and Cannabinoids (2017), supports cannabinoids as treatment for chronic pain, but highlighted the need for quality clinical trials. To fill this gap, the purpose of this study is to explore the impact of oral PEA, a non-psychoactive endocannabinoid enhancer with little to no side effects, to alter pain related biomarkers. Our central hypothesis is that PEA will alter pain related protein signatures, inflammatory markers, and neurophysiological changes in adults with KOA pain.

The investigators propose a crossover clinical trial of 20 adults with self-reported medical diagnosis of KOA and knee pain (min 4/10 on numeric rating scale). This study will explore mechanisms of taking 1200mg of oral PEA daily for seven days (loading dose) then 600 mg daily for an additional 5 weeks (six weeks total). Ten participants will take PEA for 6 weeks while the other ten will receive placebo. Then the groups will switch, with the first group receiving placebo and the second group receiving PEA. PEA takes 4 to 6 weeks to reduce KOA pain. 4,5 Participants will have blood drawn and quantitative sensory testing at baseline, 6- and 12-weeks follow-up. Participants will be asked to bring in their PEA/placebo bottles for pill counts to track adherence and will be asked about side effects at each study visit.

The investigators will test the central hypothesis and attain the objectives via the following specific aims:

Specific Aim 1: To examine the impact of oral PEA placebo on the protein signature of adults with KOA pain. We will use high-resolution liquid chromatography-tandem mass spectrometry to examine the entire proteome of the platelet rich plasma (isolated from whole blood) from each participant/time point to explore whether the PEA can alter the signaling pathways ascribed to KOA pain. We hypothesize that PEA will reduce the pro-inflammatory signaling pathways in the systemic proteome among participants in the PEA groups as compared to placebo.

Specific Aim 2: To elucidate the effects of oral PEA vs. placebo on systemic inflammatory markers related to KOA pain. We will measure key inflammatory markers in KOA including interleukin (IL)-6, IL-1β, IL-8, IL-10, IL-15, c-reactive protein (CRP) and tumor necrosis factor-α at each study visit. We hypothesize that PEA will reduce the expression of inflammatory markers seen after walking in KOA participants as compared to placebo.

Specific Aim 3: To determine the alterations in neurophysiological changes as measured by Quantitative Sensory Testing (QST) among participants taking PEA vs. placebo. For QST, we will measure the pressure pain detection and threshold, heat and cold detection and threshold, and mechanical temporal summation at the affected knee and contralateral forearm at each study visit. We hypothesize that PEA will alter central and peripheral pain pathways among adults with KOA. We will also compare the biologic pain pathways to the proteome and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 80
* English speaking
* Self reported diagnosis of osteoarthritis in one or both knees
* Self-reported average knee pain over the past month at least 4 out of 10 on a 0-10 numeric rating scale
* Agreement to abstain from all osteoarthritis pain medication (such as non-steroidal anti-inflammatory drugs or narcotics) and use only acetaminophen as a rescue medication when needed
* Can pass an evaluation to sign consent

Exclusion Criteria:

* Inflammatory arthritis (eg. Rheumatoid arthritis)
* Knee injury in past 6 months
* Knee surgery in past 12 months or total knee replacement
* Pregnant or breastfeeding
* enrolled in other knee OA rehabilitation programs or clinical trials
* Any of the following conditions: chronic kidney disease stage 3-5, unstable angina, congestive heart failure, cancer or cancer treatment (except skin)
* Oral or intra-articular glucocorticoid use in the prior 3 months; intra-articular hyaluronate use in the prior 6 months
* Opioid use in the past month
* Allergy to oat, coconut, citrus, olive, or sunflower oils, or maltodextrin

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
protein changes | 6 weeks
  we will do whole proteome sequencing from blood products to look at changes after taking PEA for 6 weeks versus placebo

SECONDARY OUTCOMES:
inflammatory markers | 6 weeks
  we will look at changes in interleukin (IL)-6, IL-1β, IL-8, IL-10, IL-15, c-reactive protein (CRP) and tumor necrosis factor-α in plasma
pain sensitivity | 6 weeks
  we will use quantitative sensitivity testing to explore changes in pain neurobiology that may occur with taking PEA versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Klinedinst, PhD, MPH, RN, Principal Investigator — University of Maryland, Baltimore; Susan Dorsey, PhD, RN, Principal Investigator — University of Maryland, Baltimore; Marc Hochberg, MD, MPH, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a preliminary study, we do not currently have a plan to share this set of data.